CLINICAL TRIAL: NCT01926834
Title: The Effect of Erigeron Injection on Acute Cerebral Infarction Serum VEGF, MMP-9 and EPC Levels
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1201/01/006284
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Cerebral Infarction
Keywords: promoting angiogenesis in multiple targets; herbal medicine; traditional chinese medicine; random clinical trial
MeSH Terms: conditions — Cerebral Infarction | interventions — Saline Solution; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Erigeron Injection (Experimental): Erigeron Injection, 30ml,qd,i.v., for 7 days
  Interventions: Drug: Erigeron Injection
- placebo (Placebo Comparator): normal saline, 500ml,i.v.,qd, for 7 days
  Interventions: Drug: placebo
- health volunteers (No Intervention): health volunteers, no drug to be given.

INTERVENTIONS:
Drug: Erigeron Injection — Erigeron Injection, 30ml, iv, qd, for 7days
  Arms: Erigeron Injection
Drug: placebo — normal saline, 500ml,i.v.,qd, for 7 days
  Other Names: normal saline, 500ml,i.v.,qd, for 7 days
  Arms: placebo

SUMMARY:
To study the effects of Erigeron Injection on human serum VEGF, MMP-9 and EPC levels after acute cerebral infarction,test is made by random double-blind controlled.patients with acute cerebral infarction were divided randomly into erigeron injection+aspirin group,aspirin group,and health people. The main indexes are the serum level of VEGF, MMP-9 and EPC.The review is made by the reference to NIHSS and so on. So, Erigeron Injection have the function of promoting angiogenesis in multiple targets through this test.

DETAILED DESCRIPTION:
OBJECTIVE:

To study the effects of Erigeron Injection on human serum VEGF, MMP-9 and EPC levels after acute cerebral infarction.

METHOD:

40 patients with acute cerebral infarction(in accordance with the inclusion criteria) were divided randomly into erigeron injection+aspirin group,aspirin group,and 20 health people. Erigeron injection+aspirin group and aspirin group drew peripheral blood on the prior treatment,the posttreatment 1th, 3th and 7th day,and tested the level of VEGF, MMP-9 and EPC.Tested the health people one time.

ELIGIBILITY:
Inclusion Criteria:

* patients aged no younger than 18yrs
* attack within 72 hours
* NIHSS score in the 2-25 points
* Ischemic Stroke occurred for the first time, or with a history of stroke disease but without sequelae
* Signed the informed consents

Exclusion Criteria:

* patients aged younger than 18yrs
* Patients with tumor, coronary heart disease, valvular heart disease, psoriasis, rheumatism, hematologic diseases, infertility, varieties of acute inflammation
* Patients with severe cognitive impairment
* Refused to cooperate or been unable to cooperation for neurological disorders
* Cerebral hemorrhage or hemorrhagic cerebral infarction
* Unstable vital signs dued to massive cerebral infarction
* Patients with serious heart, liver and renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
the serum level of VEGF,MMP-9 and EPC | 0-7days

SECONDARY OUTCOMES:
National Institute of Health of stroke scale | 0-7days

CONTACTS AND LOCATIONS:
Overall Officials: Jianwen m Guo, doctor, Principal Investigator — Guangdong Province Hospital of Tradtional Chinese Medicine